CLINICAL TRIAL: NCT01980615
Title: A Phase I, Randomized, Double-Blind Within Device, Single-Dose, Four-Period, Six-Treatment, Cross-Over Study Evaluating the Safety and Pharmacokinetics of Three Doses of Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol (BGF MDI), One Dose of Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (GFF MDI), and Two Doses of Symbicort® Inhalation Aerosol in Healthy Volunteers
Brief Title: Phase I Study Evaluating the Safety and Pharmacokinetics of Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol (BGF MDI) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT010001-00
Record Dates: First submitted 2013-10-21; First posted 2013-11-11 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- BGF MDI (PT010) Dose 1 (Experimental): BGF MDI Dose 1 taken as 2 inhalations
  Interventions: Drug: Inhaled BGF (PT010) Dose 2; Drug: Inhaled BGF (PT010) Dose 3; Drug: Inhaled GFF (PT003); Drug: Inhaled Symbicort Dose 1; Drug: Inhaled Symbicort Dose 2
- BGF MDI (PT010) Dose 2 (Experimental): BGF MDI Dose 2 taken as 2 inhalations
  Interventions: Drug: Inhaled BGF (PT010) Dose 1; Drug: Inhaled BGF (PT010) Dose 3; Drug: Inhaled GFF (PT003); Drug: Inhaled Symbicort Dose 1; Drug: Inhaled Symbicort Dose 2
- BGF MDI (PT010) Dose 3 (Experimental): BGF MDI Dose 3 taken as 2 inhalations
  Interventions: Drug: Inhaled BGF (PT010) Dose 1; Drug: Inhaled BGF (PT010) Dose 2; Drug: Inhaled GFF (PT003); Drug: Inhaled Symbicort Dose 1; Drug: Inhaled Symbicort Dose 2
- GFF MDI (PT003) (Active Comparator): GFF MDI (PT003) taken as 2 inhalations
  Interventions: Drug: Inhaled BGF (PT010) Dose 1; Drug: Inhaled BGF (PT010) Dose 2; Drug: Inhaled BGF (PT010) Dose 3; Drug: Inhaled Symbicort Dose 1; Drug: Inhaled Symbicort Dose 2
- Symbicort MDI Dose 1 (Active Comparator): Symbicort MDI taken as 2 inhalations
  Interventions: Drug: Inhaled BGF (PT010) Dose 1; Drug: Inhaled BGF (PT010) Dose 2; Drug: Inhaled BGF (PT010) Dose 3; Drug: Inhaled GFF (PT003); Drug: Inhaled Symbicort Dose 2
- Symbicort MDI Dose 2 (Active Comparator): Symbicort MDI Dose 2 taken as 2 inhalations
  Interventions: Drug: Inhaled BGF (PT010) Dose 1; Drug: Inhaled BGF (PT010) Dose 2; Drug: Inhaled BGF (PT010) Dose 3; Drug: Inhaled GFF (PT003); Drug: Inhaled Symbicort Dose 1

INTERVENTIONS:
Drug: Inhaled BGF (PT010) Dose 1
  Arms: BGF MDI (PT010) Dose 2; BGF MDI (PT010) Dose 3; GFF MDI (PT003); Symbicort MDI Dose 1; Symbicort MDI Dose 2
Drug: Inhaled BGF (PT010) Dose 2
  Arms: BGF MDI (PT010) Dose 1; BGF MDI (PT010) Dose 3; GFF MDI (PT003); Symbicort MDI Dose 1; Symbicort MDI Dose 2
Drug: Inhaled BGF (PT010) Dose 3
  Arms: BGF MDI (PT010) Dose 1; BGF MDI (PT010) Dose 2; GFF MDI (PT003); Symbicort MDI Dose 1; Symbicort MDI Dose 2
Drug: Inhaled GFF (PT003)
  Arms: BGF MDI (PT010) Dose 1; BGF MDI (PT010) Dose 2; BGF MDI (PT010) Dose 3; Symbicort MDI Dose 1; Symbicort MDI Dose 2
Drug: Inhaled Symbicort Dose 1
  Arms: BGF MDI (PT010) Dose 1; BGF MDI (PT010) Dose 2; BGF MDI (PT010) Dose 3; GFF MDI (PT003); Symbicort MDI Dose 2
Drug: Inhaled Symbicort Dose 2
  Arms: BGF MDI (PT010) Dose 1; BGF MDI (PT010) Dose 2; BGF MDI (PT010) Dose 3; GFF MDI (PT003); Symbicort MDI Dose 1

SUMMARY:
This is a Phase I, Randomized, Double-Blind Within Device, Single-Dose, Four-Period, Six-Treatment, Cross-Over Study Evaluating the Safety and Pharmacokinetics of Three Doses of Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol (BGF MDI), One Dose of Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (GFF MDI), and Two Doses of Symbicort® Inhalation Aerosol in Healthy Volunteers. The primary objective of the study is to determine a dose of budesonide that when formulated with glycopyrronium and formoterol fumarate in BGF MDI provides comparable systemic exposure [pharmacokinetics (PK)] to budesonide following administration of Symbicort MDI.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent form
* 18 and 45 years (inclusive)
* Healthy subject confirmed by a thorough medical history and physical examination, ECG, vital signs and clinical laboratory tests
* Females of childbearing potential and males with female partners of childbearing potential must agree to use medically acceptable contraception
* Body mass index (BMI) between 18.5 and 32 kg/m2 (inclusive) and a minimum weight of 50 kg at the screening visit
* Results of complete laboratory analyses should be within the normal range or determined to be not clinically significant by the Investigator

Exclusion Criteria:

* Pregnancy, nursing female subjects, or subjects trying to conceive
* Clinically significant medical conditions
* History of ECG abnormalities
* Symptomatic prostatic hypertrophy, bladder neck obstruction, or urinary retention
* Known diagnosis of glaucoma
* Known or suspected history of substance-related disorders within 1 year of screening
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) prior to screening period
* Hypersensitivity to lactose or any drug or component of the formulation(s) used in this study
* Positive screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg) or positive hepatitis C antibody at screening.
* Major surgery within four weeks or minor surgery within 2 weeks of drug administration
* Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for study participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall safety of BGF, GFF, and Symbicort MDI based on the group of outcome measures for safety. | 12 hours following study drug administration
  Safety of Three Doses of Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol (BGF MDI), One Dose of Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (GFF MDI), and Two Doses of Symbicort Inhalation Aerosol.
  The safety of BGF MDI, Symbicort MDI and GFF MDI will be assessed from physical examination findings, adverse event (AE) reporting including SAE reporting, vital signs (blood pressure, heart rate, respiratory rate and body temperature), clinical laboratory values (hematology, biochemistry, and urinalysis), and findings from 12-lead safety electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Overall pharmacokinetic profile of BGF, GFF, and Symbicort MDI based on the group of outcome measures for pharmacokinetics. | 12 hours following study drug administration
  Pharmacokinetics of Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol (BGF MDI), Symbicort MDI and GFF MDI.
  The PK of BGF MDI, Symbicort MDI and GFF MDI will be assessed and compared from plasma concentrations of each drug.
  PK parameters at all doses will include Cmax, tmax, t½, AUC0-12, AUC0-t, CL/F, Vd/F, and λz. Other PK parameters may be calculated, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics, Inc.
Locations (1):
- Pearl Therapeutics Study Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Huang Y, Assam PN, Feng C, Su R, Dorinsky P, Gillen M. Ethnic pharmacokinetic comparison of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler (BGF MDI) between Asian and Western healthy subjects. Pulm Pharmacol Ther. 2020 Oct;64:101976. doi: 10.1016/j.pupt.2020.101976. Epub 2020 Nov 2. PMID 33152467
- [Derived] Darken P, DePetrillo P, Reisner C, St Rose E, Dorinsky P. The pharmacokinetics of three doses of budesonide/glycopyrronium/formoterol fumarate dihydrate metered dose inhaler compared with active controls: A Phase I randomized, single-dose, crossover study in healthy adults. Pulm Pharmacol Ther. 2018 Jun;50:11-18. doi: 10.1016/j.pupt.2018.03.001. Epub 2018 Mar 13. PMID 29544728